CLINICAL TRIAL: NCT03966794
Title: Safety and Efficacy of Functional Neural Regeneration Collagen Scaffold Transplantation Combined With Epidural Electrical Stimulation for Spinal Cord Injury Repair
Brief Title: Functional Scaffold Transplantation Combined With Epidural Electrical Stimulation for Spinal Cord Injury Repair
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Affiliated Hospital of Logistics University of CAPF (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAS-XDA-EESCI/IGDB
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-05

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural Electrical Stimulation (Experimental)
  Interventions: Device: Epidural Electrical Stimulation
- Functional scaffold & Epidural Electrical Stimulation (Experimental)
  Interventions: Combination Product: Functional scaffold & Epidural Electrical Stimulation

INTERVENTIONS:
Device: Epidural Electrical Stimulation — Participants had finished the previous clinical trial with functional neural regeneration collagen scaffold transplantation, and will receive epidural electrical stimulation of the spinal cord in this group.
  Arms: Epidural Electrical Stimulation
Combination Product: Functional scaffold & Epidural Electrical Stimulation — Participants with acute complete SCI or chronic complete SCI will receive functional neural regeneration scaffold transplantation and epidural electrical stimulation of the spinal cord.
  Arms: Functional scaffold & Epidural Electrical Stimulation

SUMMARY:
The study is designed to assess the role of functional neural regeneration collagen scaffold transplantation combined with epidural electrical stimulation in spinal cord injury patients.

ELIGIBILITY:
Inclusion Criteria:

The enrolled participants are divided into three categories:

1. Participants had complete functional scaffold transplantation in previous study and had motor functional recovery
2. Participants With Acute Complete SCI: (1) Classification ASIA A, occurring within past 14 days; (2) Completely spinal cord injury at neurological level C4- T12/L1; (3) No serious complications
3. Participants With Chronic Complete SCI: (1) Classification ASIA A, greater than 6 months post injury and no significant further improvement within past 3 months; (2) Completely spinal cord injury at neurological level C4- T12/L1; (3) Peripheral nervous system in good condition; (4) No serious complications

Inclusion Criteria For All The Participants

1. Men or non-pregnant women, 18-60 years old
2. Ability and willingness to regular visit to hospital and follow up during the protocol Procedures
3. Accompanied by a family member
4. Signed informed consent

Exclusion Criteria:

1. Obvious muscle atrophy or fibrosis
2. Decline in peripheral nerve function
3. A current diagnosis of diseases affecting spinal cord injury recovery or rehabilitation training (e.g., brain injury, cerebral hemorrhage, cognitive impairment, other central nervous system diseases)
4. Having serious health problems, (e.g., cardiovascular disease, diabetes, autoimmune diseases, tumors or severe hypertension) or serious complications (e.g. severe bedsores, pulmonary infection, respiratory disorders)
5. Pregnancy or lactation
6. History of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders
7. No family member accompany or can not get in touch with family members
8. Poor compliance, difficult to complete the study
9. Any other conditions that might increase the risk of participants or interfere with the clinical trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability assessed by Adverse Events | Up to 6 months
  Proportion of patients with postoperative infections and serious adverse events (SAEs) will be assessed by long term follow-up
Change in ASIA Impairment Scale | Baseline, 1, 3 , 6, 12 and 24 months post-treatment
  American Spinal Injury Association Impairment Scale of A, B, C, D or E will be assessed before and after transplantation.

SECONDARY OUTCOMES:
Change in ASIA motor score | Baseline, 1, 3 , 6, 12 and 24 months post-treatment
Change in Functional Independence Measure (FIM) | Baseline, 1, 3 , 6, 12 and 24 months post-treatment
Change in Somatosensory Evoked Potentials (SSEP) monitoring | Baseline, 1, 3 , 6, 12 and 24 months post-treatment
Change in Motor Evoked Potentials (MEP) monitoring | Baseline, 1, 3 , 6, 12 and 24 months post-treatment
Changes at the Transplantation Site in Spinal Cord by Magnetic Resonance Imaging (MRI) | Baseline, 1, 3 , 6, 12 and 24 months post-treatment
Change in Walking Speed | Baseline, 1, 3 , 6, 12 and 24 months post-treatment
Change in Stride length | Baseline, 1, 3 , 6, 12 and 24 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- Affiliated Hospital of Logistics Universtiy of CAPF, Tianjin, China